CLINICAL TRIAL: NCT06832930
Title: A Real-World Case Study Evaluating the Efficacy and Safety of Bronchial Navigation Localization Device-Assisted Cryobiopsy
Brief Title: A Real-World Case Study Evaluating the Efficacy and Safety of RBS Cryobiopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, professor, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBS-cryobiopsy
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Pulmonary Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RBS group (Experimental): Patients in RBS group would undergo cryobiopsy with the help of RBS
  Interventions: Procedure: unicorn robotic bronchoscopy system
- Control group (Other): Patients in control group would undergo cryobiopsy with the help of conventional navigation technology.
  Interventions: Procedure: Conventional navigation bronchoscopy

INTERVENTIONS:
Procedure: unicorn robotic bronchoscopy system — cryobiopsy with the help of robotic bronchoscopy system
  Arms: RBS group
Procedure: Conventional navigation bronchoscopy — cryobiopsy with the help of Conventional navigation bronchoscopy
  Arms: Control group

SUMMARY:
The goal of this clinical trial is tois to assess the effectiveness and safety of RBS (Robotic Bronchoscopy System)-assisted cryobiopsy in real-world clinical settings in adult patients (aged ≥18 years) with suspected pulmonary lesions requiring diagnostic bronchoscopic evaluation. The main questions it aims to answer are:

Does RBS-assisted cryobiopsy improve diagnostic yield compared to conventional non-RBS-guided cryobiopsy? Is RBS-assisted cryobiopsy associated with a lower incidence of procedure-related complications (e.g., bleeding, pneumothorax) compared to conventional methods? Researchers will compare the RBS group (patients undergoing RBS-assisted cryobiopsy) with the control group (patients undergoing cryobiopsy with conventional navigation techniques, such as ENB, VBN) to evaluate differences in diagnostic accuracy and safety outcomes.

Participants will:

Provide informed consent for bronchoscopic cryobiopsy. Undergo pre-procedure imaging and clinical evaluation. Receive either RBS-assisted or conventional cryobiopsy based on clinical indication and operator discretion.

Be monitored for immediate and delayed complications .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Patients are eligible for inclusion if they meet all of the following criteria:

  1. Age ≥18 years and ≤75 years, with no gender restrictions;
  2. Presence of a peripheral lung lesion on chest CT
  3. Patients voluntarily agree to undergo bronchoscopy and meet the requirements for the procedure;
  4. patients are capable of understanding the purpose of the trial, demonstrate good compliance with the examinations and follow-up, voluntarily participate in the clinical trial, and sign an informed consent form.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from this study:

  1. Presence of contraindications for bronchoscopy, including: active massive hemoptysis; recent myocardial infarction or unstable angina; severe cardiac or pulmonary dysfunction; severe hypertension and arrhythmias; uncorrectable bleeding tendencies or severe coagulation disorders (such as platelet count <60×10^9/L), uremia; severe pulmonary artery hypertension; severe superior vena cava syndrome; intracranial hypertension; acute cerebrovascular events; aortic dissection or aneurysm; multiple bullae; extreme systemic exhaustion;
  2. Female patients who are breastfeeding, pregnant, or planning pregnancy;
  3. Patients with electromagnetic active implantable medical devices;
  4. Subjects allergic to anesthetics; or with a history of multiple severe allergies, hereditary allergy history;
  5. Those who have participated in or are currently participating in drug clinical trials within 3 months before screening, or have participated in other medical device clinical trials within 30 days;
  6. Any other conditions deemed unsuitable for participation in this clinical trial by the investigator.

     Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
overall diagnostic yield | 6 months after biopsy
  Overall diagnostic yield was considered as the primary outcome, defined as the number of cases in which the diagnosis of bronchoscopy matched the final diagnosis, divided by the total number of completed cases during follow-up. A lesion was considered malignant if tumor cells were found in histological and/or cytological specimens. It was considered benign if pathological evaluation showed specific benign pathology and/or non-specific benign lesions confirmed by MDT discussion.

SECONDARY OUTCOMES:
Navigation success rate | During the bronchoscopy
  The success rate of navigation = (the number of lesions judged as successfully navigated / the total number of lesions undergoing transbronchial lung biopsy) * 100%. The criteria for judging successful navigation: if the lesion edge is confirmed by imaging equipment and the researcher deems it feasible for biopsy, it is considered a successful navigation; otherwise, it is regarded as a failed navigation. For those with a clear diagnosis through the research procedure, all are considered successful navigation.

REFERENCES:
- [Background] de Baere T, Woodrum D, Tselikas L, Abtin F, Littrup P, Deschamps F, Suh R, Aoun HD, Callstrom M. The ECLIPSE Study: Efficacy of Cryoablation on Metastatic Lung Tumors With a 5-Year Follow-Up. J Thorac Oncol. 2021 Nov;16(11):1840-1849. doi: 10.1016/j.jtho.2021.07.021. Epub 2021 Aug 9. PMID 34384914